CLINICAL TRIAL: NCT04454684
Title: An Open-Label, Multi-Site Phase 2 Study of the Safety and Feasibility of MDMA-Assisted Psychotherapy for Eating Disorders
Brief Title: A Multi-Site Study of MDMA-Assisted Psychotherapy for Eating Disorders
Acronym: MED1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No site was initiated.
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED1
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Anorexia Nervosa Restricting Type; Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Examining safety and effects of three sessions of MDMA-assisted psychotherapy
Masking Description: This study will be open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AN-R: MDMA-assisted Psychotherapy (Experimental): Three Experimental Sessions of MDMA-assisted psychotherapy. The first Experimental Session involves 80mg midomafetamine HCl followed by a supplemental half-dose of 40 mg midomafetamine HCl 1.5 to 2 hours later, unless contraindicated. The second and third Experimental Sessions involve a flexible dose of 80 or 120 mg midomafetamine HCl followed by a supplemental half-dose of 40 or 80 mg midomafetamine HCl, respectively, 1.5 to 2 hours later, unless contraindicated.
  Interventions: Drug: Midomafetamine; Behavioral: Non-directive therapy; Behavioral: Therapy
- BED: MDMA-assisted Psychotherapy (Experimental): Three Experimental Sessions of MDMA-assisted psychotherapy. The first Experimental Session involves 80mg midomafetamine HCl followed by a supplemental half-dose of 40 mg midomafetamine HCl 1.5 to 2 hours later, unless contraindicated. The second and third Experimental Sessions involve a flexible dose of 80 or 120 mg of midomafetamine HCl followed by a supplemental half-dose of 40 or 80 mg midomafetamine HCl, respectively, 1.5 to 2 hours later, unless contraindicated.
  Interventions: Drug: Midomafetamine; Behavioral: Non-directive therapy; Behavioral: Therapy
- Caregivers: Psychotherapy (Experimental): Psychotherapy alone
  Interventions: Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine — Initial dose of 80 or 120 mg midomafetamine HCl administered orally at the start of each of three psychotherapy sessions, followed by a supplemental half-dose of 40 to 60 mg midomafetamine HCl 1.5 to 2.5 hours later, unless contraindicated.
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine HCl
  Arms: AN-R: MDMA-assisted Psychotherapy; BED: MDMA-assisted Psychotherapy
Behavioral: Non-directive therapy — Non-directive therapy will be conducted during Experimental Sessions.
  Other Names: Manualized MDMA-assisted therapy
  Arms: AN-R: MDMA-assisted Psychotherapy; BED: MDMA-assisted Psychotherapy
Behavioral: Therapy — Therapy will be conducted during Preparatory Sessions and Integrative Sessions.

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy and caregiver involvement are safe and effective in treating female participants with eating disorders.

The main question it aims to answer is: Does MDMA-assisted therapy reduce eating disorder symptoms?

Participants will undergo two non-drug preparatory therapy sessions and their caregiver will undergo one non-drug preparatory therapy session. Participants will undergo three sessions of MDMA-assisted therapy followed by non-drug integrative therapy sessions alone as well as together with their caregiver.

DETAILED DESCRIPTION:
This Phase 2, open-label, multi-site study will explore the safety and feasibility MDMA-assisted psychotherapy and adjunctive caregiver involvement in the treatment of 18 participants with eating disorders. The study will enroll 12 participants with anorexia nervosa restricting-type (AN-R) and six participants with binge eating disorder (BED). A supportive caregiver, such as a parent or partner, for each participant will also be recruited to participate in the study and receive non-drug psychotherapy support.

The study will consist of two Preparatory Sessions for each participant with an eating disorder and one Preparatory Session for each caregiver participant. During the treatment period, participants with eating disorders will undergo three Experimental Sessions of MDMA-assisted psychotherapy, lasting approximately eight hours each. The first Experimental Session will be followed by Individual Integrative Sessions for the participant with an eating disorder and caregiver participant separately as well as a combined Dyadic Integrative Session with both the participant with an eating disorder and their caregiver together. After the second and third Experimental Session, just the participant with an eating disorder will have an Individual Integrative Session before the combined Dyadic Integrative Session with their caregiver.

The first Experimental Session will involve a dose of 80 mg midomafetamine HCl, followed by a supplemental half-dose of 40 mg 1.5 to 2 hours later, unless contraindicated. The second and third Experimental Sessions will involve a flexible dose of 80 or 120 mg of midomafetamine HCl, followed by a supplement half-dose of 40 or 60 mg, respectively, unless contraindicated. The primary outcome measure is the change in Eating Disorder Examination (EDE) results at Baseline to Visit 16 (Study Termination).

ELIGIBILITY:
Inclusion Criteria for Eating Disorder (ED) Participants:

* Are 21 to 65 years old.
* Are assigned female at birth.
* Are fluent in speaking and reading the English language and can provide written informed consent.
* Are able to swallow pills.
* Agree to have study visits recorded to audio and video.
* Are willing to include a consenting caregiver as a co-participant in elements of the study with whom the study team will have regular contact. This person must be willing and able to be reached by the investigators in case of emergency.
* If connected to a psychotherapist at the time of recruitment into the study, participants may not change therapists, change the frequency of therapy, or commence any new type of therapy until after the Study Termination Visit, 1 month after the final Experimental Session.
* Have an identified Primary Care Physician (PCP) and provide consent for the investigator to communicate with PCP, as needed.
* If AN-R diagnosis, are currently participating in a recognized ED treatment program.
* Are willing to sign a release for the investigators to communicate directly with their therapist, physician if relevant, as well treatment providers where they were currently or previously engaged an ED-specific episode of treatment.
* Live within reasonable driving distance of the study site (equal to or less than an estimated 2-hour drive from the study site).
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control
* Agree to inform the investigators within 48 hours of any medical conditions and procedures.
* Agree to lifestyle modifications, comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not participate in any other interventional clinical trials during the duration of the study, remain overnight at the study site (or appropriate location approved by the research team) after each Experimental Session, not operate a vehicle within 24 hours after MDMA administration, and commit to medication dosing, therapy, and study procedures.
* Have Anorexia Nervosa, Restricting Type or Binge Eating Disorder.
* Current or past treatment were not successful to retain remission
* Have a BMI > 15 kg/m2 and are medically stable according to screening Electrocardiogram (ECG), blood pressure monitoring, and blood and urine laboratory screening results.

Exclusion Criteria for Eating Disorder (ED) Participants:

* Are not able to give adequate informed consent.
* Have any current problem which, in the opinion of the investigator or Medical Monitor, might interfere with participation.
* Cannot identify a supportive caregiver to participate in the study (or the caregiver does not meet eligibility criteria).
* Have a blood or needle phobia that interferes with obtaining necessary blood work
* Have a history of significant medical disorders
* Have any current problematic patterns of alcohol or other substance use
* Require use of prohibited concomitant medications for this study, including those that prolong the QT/QTc interval during Experimental Sessions.
* Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate.
* Have uncontrolled hypertension or history of ventricular arrhythmia.
* Have Wolff-Parkinson-White syndrome or any other accessory pathway.
* Have a marked Baseline prolongation of QTcF interval (e.g., repeated demonstration of a QTcF interval > 450 ms).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have symptomatic liver disease.
* Have a history of non-ED-symptom-related hyponatremia or hyperthermia.
* Are pregnant or nursing, or are persons of childbearing potential who are not practicing (or not willing to practice) an effective means of birth control.
* Are assessed to be medically unstable

Inclusion Criteria for Caregiver (CG) Participants:

* Are fluent in speaking and reading the English language and can provide written informed consent.
* Are at least 18 years old.
* Are the parent, partner, or other significant caregiver of the ED Participant.
* Are involved in caregiving at least 2 hours a week (i.e. companionship, meal support, emotional support, driving to appointments, financial support, etc.).
* Are willing to provide their loved one with meal/symptom support and emotional support throughout the study.
* Live within reasonable driving distance of the study site
* If in ongoing psychotherapy at the time participants are recruited into the study, caregiver participants may continue to see their outside therapist during the course of the study. Caregiver participants must sign a release for the investigators to communicate directly with their therapist. CG Participants may not change therapists, increase the frequency of therapy, or commence any new type of therapy until after their Study Termination Visit.
* Are willing to commit to Preparatory and Integrative Sessions, completion of evaluation instruments and other study procedures, and being contacted for all necessary telephone contacts.
* Agree to have study visits recorded to audio and video.

Exclusion Criteria for Caregiver (CG) Participants:

* Have a current eating disorder.
* Are unable to give adequate informed consent.
* Report any current problem which in the opinion of the investigator or Medical Monitor might interfere with enrollment or ongoing participation.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 0 (Actual)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Examination Interview (EDE) Global Score from Baseline to Visit 16 (Study Termination) | Baseline to 17 weeks post-enrollment
  The Eating Disorder Examination Interview (EDE) is a semi-structured interview that assesses the frequency of key behavioral features of eating disorders as well as the severity of specific ED psychopathology. The EDE is widely considered to be the gold standard for assessing eating disorder pathology and can detect differences between individuals with anorexia nervosa and binge eating disorder.
  The EDE consists of four subscales: Restraint, Eating Concern, Shape Concern, and Weight Concern. The interview rates each question based on its frequency in the past month from a score of 0 (feature not present) to 6 (feature present every day). Subscale scores are calculated by totaling the scores in each subscale and dividing by the total number of items in the subscale. The overall or global score is calculated by summing the four subscale scores and dividing by four. The higher the score, the greater the eating disorder severity and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Lafrance, PhD, Principal Investigator — Emotion Science

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available wehn all participants have completed the study.
Access Criteria: Interested persons should correspond with the central contact for the multi-site study.

REFERENCES:
- [Background] Cooper, Z. and C. Fairburn, The eating disorder examination: A semi-structured interview for the assessment of the specific psychopathology of eating disorders. International journal of eating disorders, 1987. 6(1): p. 1-8.
- [Background] Fairburn, C., Z. Cooper, and M. O'Connor, Eating Disorder Examination (Edition 17.0D; April, 2014). 2014: https://www.corc.uk.net/media/1951/ede_170d.pdf.
- [Background] Keel PK, Brown TA. Update on course and outcome in eating disorders. Int J Eat Disord. 2010 Apr;43(3):195-204. doi: 10.1002/eat.20810. PMID 20186717